CLINICAL TRIAL: NCT05035303
Title: Can Trajectory Nor-epinephrine Infiltration Reduce Blood Loss During Percutaneous Nephrolithotomy?: A Double-blind Randomized Placebo Controlled Study.
Brief Title: Can Trajectory Nor-epinephrine Infiltration Reduce Blood Loss During Percutaneous Nephrolithotomy (PCNL)?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Associate professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RC-200310
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double- blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nor-Epinephrine (NE)-Group (Active Comparator): The PCNL tract is infiltrated by Nor-Epinephrine before its dilatation.
  Interventions: Procedure: Nor-Epinephrine injection versus saline during PCNL
- S-Group (Placebo Comparator): The PCNL tract is infiltrated by Normal Saline before its dilatation.
  Interventions: Procedure: Nor-Epinephrine injection versus saline during PCNL

INTERVENTIONS:
Procedure: Nor-Epinephrine injection versus saline during PCNL — The PCNL tract is infiltrated by Nor-Epinephrine or Normal Saline before its dilatation.

SUMMARY:
during PCNL; A few milliliters of nor-epinephrine is injected into the intended tract after puncture of pelvicalyceal system and before its dilatation compared to injection of saline (placebo). hemoglobin change & blood loss is estimated and will compared.

DETAILED DESCRIPTION:
All patients of are positioned in lithotomy position and 6 F open tip ureteral catheter is fixed by cystoscope. Then, A pelvicalyceal system is punctured under ultrasound and/or fluoroscopic guidance, then a 18 Gauge (G) puncture needle is introduced toward the desired calyx and a 0.038 inch guide wire is inserted. then 20 G Chiba needle is introduced alongside the puncture needle for infiltration of the whole tract by either a few milliliters of nor-epinephrine or saline. then, the tract is dilated over the guide wire, lastly an Amplatz sheath was inserted.

nephroscope is used for stones disintegration by pneumatic or laser lithotripter . Fragments are washed out or removed by forceps.

ELIGIBILITY:
Inclusion Criteria:

* renal stones>2 cm

Exclusion Criteria:

* coagulopathy, congenital anomalies, active Urinary tract infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
hemoglobin drop | 72 hours post intervention
  the lower drop is better
blood loss | immediately after surgery
  the lower loss is better

SECONDARY OUTCOMES:
stone free rate | within 3 months post-operative
  the higher is better
adverse events | within 30 days post-operative
  the lower is better

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Shaer, Principal Investigator — Faculty of medicine, Banha university
Locations (2):
- Egypt (2):
  - Banha University Hospitals, Banhā, Kalubiaya
  - Banha university hospital, Banhā, Qalyubia Governorate

IPD SHARING:
Plan to Share IPD: No